CLINICAL TRIAL: NCT04898595
Title: Discontinuation of Continuous Renal Replacement Therapy in Patients with Acute Kidney Injury: a Pilot Quasi-experimental Study (DC-CRRT)
Brief Title: Discontinuing CRRT in Patients with Acute Kidney Injury
Acronym: DC-CRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Khaled Shawwa, Assistant Professor, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2101226767
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: This is a prospective quasi-experimental (before-after) study of patients with acute kidney injury requiring continuous renal replacement therapy in the intensive care unit. This will be a quasi-experimental study design due to the nature of the intervention and the processes of care leading to making a clinical decision. Patients with AKI on CRRT will be prospectively recruited. Patients recruited during the first half of the study will be in the control arm where usual process of care will not be altered. After accrual, patients recruited for the second half will receive the intervention where discontinuation of CRRT will be guided by a set of criteria based on the patient's hemodynamic status and other factors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Process of Care (No Intervention): No intervention
- Standardized approach to discontinuation of CRRT (Experimental): Criteria-driven approach
  Interventions: Procedure: Discontinuation of CRRT

INTERVENTIONS:
Procedure: Discontinuation of CRRT — Discontinuation of CRRT will be guided by an algorithm based on patient current condition.
  Arms: Standardized approach to discontinuation of CRRT

SUMMARY:
In this study, investigators are going to test whether a standardize approach to discontinuation of Continuous Renal Replacement Therapy (CRRT) using a set of criteria improves outcomes. These criteria are based on the best available evidence. In a systematic review, aside from urine output, there was no one factor that predicted successful weaning of RRT in patients with AKI. Urine output prior to discontinuation of RRT was the most commonly described and robust predictor. The pooled analysis found a sensitivity of 66.2% and specificity of 73.6% for urine output to predict successful RRT discontinuation. Patients with AKI on CRRT recruited during the first half of the study will be controls (usual process of care). After accrual, patients recruited for the second half will receive the intervention where discontinuation of CRRT will be guided by a set of criteria based on the patient's hemodynamic status and other factors.

DETAILED DESCRIPTION:
To the investigator's knowledge, no study has evaluated the impact of a standardized approach to de-escalation of Continuous Renal Replacement Therapy (CRRT) in patients with AKI. Exposure to more frequent and higher intensity RRT has been associated with delayed renal recovery. There is scant evidence in the literature on benefit or harm associated with a standardized approach to de-escalation of CRRT on the outcomes of successful weaning of CRRT, impact on CRRT duration, renal recovery, safety and adverse events. Thus, this generates a clinical equipoise. Therefore, this study should help guide nephrologists and intensivists on the appropriate management of CRRT in patients with AKI.

This is a prospective quasi-experimental (before-after) study of patients with acute kidney injury requiring continuous renal replacement therapy in the intensive care unit. It will be based on Good Clinical Practice Standards and performed under IRB supervision. This will be a quasi-experimental study design due to the nature of the intervention and the processes of care leading to making a clinical decision. Patients with AKI on CRRT will be prospectively recruited. Patients recruited during the first half of the study will be in the control arm where usual process of care will not be altered. After accrual, patients recruited for the second half will receive the intervention where discontinuation of CRRT will be guided by a set of criteria based on the patient's hemodynamic status and other factors. A decision tree form would be filled by one of the team members each day. This will increase adherence to the protocol and allow us to track reasons for not discontinuing CRRT when it is suggested to do so.

Patients will be approached within 24-36 hours of starting CRRT. Patients will be eligible for trial entry after the decision is made to pursue CRRT. Patients with provided informed consent will be accrued in the study.

The hypothesis is that the intervention arm will lead to earlier discontinuation of CRRT. This may translate to less treatment-associated adverse events, namely intradialytic hypotension, and potentially improve the chance of renal recovery. Investigators will collect data on persistent kidney dysfunction at 30 days after AKI as defined by persistent need for RRT or doubling of baseline creatinine.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of acute kidney injury
* Being started on continuous renal replacement therapy

Exclusion criteria:

* Diagnosis of chronic kidney disease stage 5 or end-stage renal disease
* Having received a kidney transplant
* Moribund patients (who are expected to die within 1 day of CRRT initiation)
* Presence of an intoxication requiring extracorporeal removal
* RRT within the previous 1 month
* Rapidly progressive glomerulonephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Successful discontinuation of Continuous Renal Replacement Therapy | 7 consecutive days post last CRRT performed
  Successful discontinuation of CRRT is defined by being free from any form of renal replacement therapy for at least 7 consecutive days. We will measure the difference in the proportion of participants who achieve successful discontinuation of CRRT between the two groups.

SECONDARY OUTCOMES:
Major adverse kidney events (MAKE30) | Up to 30 days
  The composite outcome of death, continued need of dialysis, and persistent kidney dysfunction (defined as doubling of baseline creatinine) at day 30 after starting CRRT.
CRRT duration | 1 to 100 days
  Absolute number of days the subject received CRRT prior to first discontinuation.
Intermittent hemodialysis after CRRT discontinuation | Within 7 days post DC CRRT
  Number of subjects that require intermittent hemodialysis after discontinuation of CRRT
Adverse events occurring within 7 days after discontinuation of CRRT | Within 7 days post DC CRRT
  Any adverse events, from the below list, that occur within 7 days after discontinuation of CRRT
  * Hyperkalemia with potassium of >6.1 mmol/L
  * Severe metabolic acidosis (defined as pH ≤7·20, PaCO2 ≤45 mm Hg, and bicarbonate concentration ≤20 mmol/L)
  * Complications of hypervolemia
  * Catheter-related blood stream infections

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Shawwa, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No